CLINICAL TRIAL: NCT03585244
Title: A Study to Assess Change in Weight Over Six Months in Prader-Willi Syndrome
Brief Title: Weight Change in PWS Over Six Months
Status: Completed | Type: Observational
Sponsor: Foundation for Prader-Willi Research (Other)
Collaborators: Prader-Willi Syndrome Association USA (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_WS
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Weight Change, Body
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Prader-Willi Syndrome: Individuals with Prader-Willi Syndrome aged 12 and over will be recruited to gather data on weekly weight over six months
  Interventions: Other: weekly weight

INTERVENTIONS:
Other: weekly weight — weekly weight data collection for six months

SUMMARY:
This is a completely text-messaging based study and all data will be collected via surveys administered on a mobile phone. For this study, we will gather and analyze data on changes in body weight over a 6-month interval in individuals aged 12 and over. This will help us learn more about the normal variation in weight, over time, in the PWS population.

DETAILED DESCRIPTION:
The incidence and natural history of several PWS symptoms are poorly defined. In this text-messaging based study we will gather and analyze data on changes in body weight over a 6-month interval, in individuals aged 12 and over. We would like to learn about the normal weight variation in the PWS population.

We anticipate that this study will inform future clinical trials for hyperphagia/obesity related therapies, and provide a basis for understanding how well potential therapies are working. For this study, there will be no intervention and the all data will be collected via texting.

ELIGIBILITY:
Inclusion Criteria:

Participants with PWS are eligible for this study. Eligible PWS participants must be 12 years and older. Participant/legal representative of participant must have a text messaging enabled mobile phone in order to participate in the study Participants must reside in the U.S. or Canada

-

Exclusion Criteria:

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with PWS
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Remote, Walnut, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individuals With Prader-Willi Syndrome
Started | 180
Completed | 165
Not Completed | 15
Not completed — Withdrawal by Subject | 15

BASELINE CHARACTERISTICS:
Arm/Group | Individuals With Prader-Willi Syndrome
Number analyzed (Participants) | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 88
  Between 18 and 65 years | 77
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 84
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 150
  Canada | 15
Weight [Mean (Standard Deviation); unit: Kilograms] | 76.8 (30.7)
Height [Mean (Standard Deviation); unit: Centimeters] | 157.2 (13.2)
BMI [Median (Full Range); unit: Kilograms/m^2] | 28.6 [13.2 to 88.0]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Change in Weight
Description: weekly weight data will be collected via text for 6 months
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: Percent of change in weight
Arm/Group | Individuals With Prader-Willi Syndrome
Number analyzed (Participants) | 165
Percent of change in weight | 2.35 (5.3)

2. Primary Outcome: Percent of Change in BMI
Description: weekly weight and height data will be collected via text for 6 months
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: Percent of change in BMI
Arm/Group | Individuals With Prader-Willi Syndrome
Number analyzed (Participants) | 165
Percent of change in BMI | 1.42 (5.9)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Individuals With Prader-Willi Syndrome
All-Cause Mortality (participants affected / at risk) | 0/165
Serious Adverse Events (participants affected / at risk) | 0/165
Other Adverse Events (participants affected / at risk) | 0/165

LIMITATIONS AND CAVEATS:
This study was all text message based data collection so we were only able to collect limited information and did not collect race or ethnicity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03585244/Prot_000.pdf